CLINICAL TRIAL: NCT03195517
Title: Effects of a 3-month Weight-bearing and Resistance Exercise Training on Circulating Osteoprogenitor Cells and Bone Formation Markers in Postmenopausal Women With Low Bone Mass.
Brief Title: Effects of Physical Training on Bone Turnover and Quality of Life in Osteopenic Postmenopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Rita Lombardini, Principal Investigator, University Of Perugia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OPCuriamo-1
Record Dates: First submitted 2017-06-15; First posted 2017-06-22 (Actual); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Osteopenia; Bone Turnover Markers; Quality of Life
Keywords: Osteopenia; Physical activity; Bone turnover markers; Osteoprogenitor cells; Quality of life
MeSH Terms: conditions — Bone Diseases, Metabolic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This was an interventional, single group assignment study in which the subjects were first assigned to the control group and, after 1-month interval with no physical training, were shifted into the 3-months exercise intervention group. Thus, the subjects acted as their own control at the end of the study.

ARMS (2):
- Physical Exercise (Experimental): The exercise program was performed at C.U.R.I.A.Mo. Institute of "Università degli Studi di Perugia". Twenty-four exercise sessions were provided, carried out twice a week for three months. Each session was supervised by two graduated trainers and two medical doctors with a maximum attendance of 5 patient/group.
  Each session lasted 45 minutes divided into 15 minutes of aerobic activity and 30 minutes of weight-bearing and resistance activities.
  This latter section was specifically projected for adults and older adults with increased risk of fractures and was intended to improve muscle strength and flexibility, balance and, as a result, to prevent the risk of falls.
  Interventions: Other: Physical exercise
- No additional physical exercise (No Intervention): Usual recommendations for prevention of fractures in adults and elderly.

INTERVENTIONS:
Other: Physical exercise
  Arms: Physical Exercise

SUMMARY:
The aim of our research was to define both in vivo and in vitro whether and to what extent an high-impact exercise program would affect bone cell turnover and improve the QoL in osteopenic postmenopausal women.

DETAILED DESCRIPTION:
Subjects were selected among those attending the "Bone and Mineral Metabolism Disorders" Clinic of Perugia University, Italy, since May 2nd 2015 and January 31st 2016. A total of 33 post-menopausal women volunteered to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* bone mineral density T-score less than -1 but more than -2.5 in the total hip or lumbar spine (L1-L4) by dual energy x-ray absorptiometry
* be able to attend an exercise program 2 times per week over the 3-month period
* stated availability throughout the entire study period

Exclusion Criteria:

* secondary causes of bone loss such as osteomalacia, glucocorticoid medication
* co-morbidities that would interfere with participation in exercise such as severe heart or pulmonary disease, inflammatory joint disease, severe osteoarthritis, psychiatric condition
* physical or orthopaedic disabilities that would place the subject at risk or limit their ability to perform exercise
* a past vertebral fracture
* history of chronic diseases, such as renal, hepatic, cardiac, and rheumatic diseases
* current or prior use of drugs that could interfere with bone mass (i.e. glucocorticoids, antiresorptive drugs and hormonal replacement therapy)

Ages: 52 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lombardini, Principal Investigator — University Of Perugia

REFERENCES:
- [Background] Turner CH, Robling AG. Mechanisms by which exercise improves bone strength. J Bone Miner Metab. 2005;23 Suppl:16-22. doi: 10.1007/BF03026318. PMID 15984409
- [Background] Pasqualini L, Leli C, Ministrini S, Schillaci G, Zappavigna RM, Lombardini R, Scarponi AM, Mannarino E. Relationships between global physical activity and bone mineral density in a group of male and female students. J Sports Med Phys Fitness. 2017 Mar;57(3):238-243. doi: 10.23736/S0022-4707.16.06054-0. Epub 2016 May 31. PMID 27244129
- [Background] Martyn-St James M, Carroll S. A meta-analysis of impact exercise on postmenopausal bone loss: the case for mixed loading exercise programmes. Br J Sports Med. 2009 Dec;43(12):898-908. doi: 10.1136/bjsm.2008.052704. Epub 2008 Nov 3. PMID 18981037
- [Background] Robling AG, Niziolek PJ, Baldridge LA, Condon KW, Allen MR, Alam I, Mantila SM, Gluhak-Heinrich J, Bellido TM, Harris SE, Turner CH. Mechanical stimulation of bone in vivo reduces osteocyte expression of Sost/sclerostin. J Biol Chem. 2008 Feb 29;283(9):5866-75. doi: 10.1074/jbc.M705092200. Epub 2007 Dec 17. PMID 18089564
- [Background] Li WC, Chen YC, Yang RS, Tsauo JY. Effects of exercise programmes on quality of life in osteoporotic and osteopenic postmenopausal women: a systematic review and meta-analysis. Clin Rehabil. 2009 Oct;23(10):888-96. doi: 10.1177/0269215509339002. Epub 2009 Aug 28. PMID 19717503
- [Background] Pirro M, Leli C, Fabbriciani G, Manfredelli MR, Callarelli L, Bagaglia F, Scarponi AM, Mannarino E. Association between circulating osteoprogenitor cell numbers and bone mineral density in postmenopausal osteoporosis. Osteoporos Int. 2010 Feb;21(2):297-306. doi: 10.1007/s00198-009-0968-0. Epub 2009 May 30. PMID 19484167
- [Background] Lips P, Leplege A (2000). Development and validation of quality of life questionnaire for patients with vertebral fractures: Qualeffo-41. Quality of Life Research 9(6a):763-766.
- [Background] Adami S, Gatti D, Viapiana O, Fiore CE, Nuti R, Luisetto G, Ponte M, Rossini M; BONTURNO Study Group. Physical activity and bone turnover markers: a cross-sectional and a longitudinal study. Calcif Tissue Int. 2008 Dec;83(6):388-92. doi: 10.1007/s00223-008-9184-8. Epub 2008 Oct 24. PMID 18949504
- [Derived] Pasqualini L, Ministrini S, Lombardini R, Bagaglia F, Paltriccia R, Pippi R, Collebrusco L, Reginato E, Sbroma Tomaro E, Marini E, D'Abbondanza M, Scarponi AM, De Feo P, Pirro M. Effects of a 3-month weight-bearing and resistance exercise training on circulating osteogenic cells and bone formation markers in postmenopausal women with low bone mass. Osteoporos Int. 2019 Apr;30(4):797-806. doi: 10.1007/s00198-019-04908-9. Epub 2019 Feb 26. PMID 30809725

RESULTS

PARTICIPANT FLOW:
Groups:
- Control/Exercise Training: At the start of the study, all participants were assigned to 1-month non-exercise control group. Measurements of bone formation markers, circulating osteoprogenitor cells and health-related quality of life were evaluated at the time of enrollment and after 1 month run-in.
  All study participants, assigned to 1-month non-exercise control group, were shifted into the exercise intervention group. Measurements of bone formation markers, circulating osteoprogenitor cells, physical fitness and health-related quality of life were evaluated after 3-months of high-impact exercise training.
Period: Overall Study
Arm/Group | Control/Exercise Training
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Control/Exercise Training: 33 osteopenic postmenopausal women were included in the study. Bone formation markers, circulating osteoprogenitor cells and health-related quality of life were evaluated at the time of enrollment, after 1 month run-in and after 3 months of high-impact exercise training.
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 12
Age, Customized [Mean (Standard Deviation); unit: years] | 62.6 (5.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 33

OUTCOME MEASURES:

1. Primary Outcome: Variation in Serum Levels of Procollagen 1 N-terminal Peptide (P1NP)
Description: P1NP is the most reliable serum marker of bone formation commercially available at the moment
Time Frame: Baseline - Week 4
Population: Post-menopausal women with low bone mass at dual energy X-ray absorptiometry (DEXA) measurement, compatible with osteopenia (T-score between -1 DS and -2.5 DS)
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | No Additional Physical Exercise
Number analyzed (Participants) | 33
mcg/L
  P1NP, Baseline | 58.34 (9.24)
  P1NP, W4 | 57.91 (8.49)
Statistical Analysis 1: Comparison: No Additional Physical Exercise; Test type: Other; p = 0.05, t-test, 1 sided

2. Primary Outcome: Variation in Serum Levels of Procollagen 1 N-terminal Peptide (P1NP).
Description: P1NP is the most reliable serum marker of bone formation, commercially available at the moment.
Time Frame: Week 4 - Week 12
Population: Post-menopausal women with low bone mass at DEXA measurement, compatible with osteopenia (T-score between -1 DS and -2.5 DS)
Measure: Mean (Standard Deviation); unit: mcg/L
Groups:
- Physical Exercise: The exercise program was performed at C.U.R.I.A.Mo. Institute of "Università degli Studi di Perugia". Twenty-four exercise sessions were provided, carried out twice a week for three months. Each session was supervised by two graduated trainers and two medical doctors with a maximum attendance of 5 patient/group.
  Each session lasted 45 minutes divided into 15 minutes of aerobic activity and 30 minutes of weight-bearing and resistance activities.
  This latter section was specifically projected for adults and older adults with increased risk of fractures and was intended to improve muscle strength and flexibility, balance and, as a result, to prevent the risk of falls.
  Physical exercise
Arm/Group | Physical Exercise
Number analyzed (Participants) | 33
mcg/L
  P1NP, W4 | 57.91 (8.49)
  P1NP, W12 | 64.87 (12.67)
Statistical Analysis 1: Comparison: Physical Exercise; Test type: Other; p = 0.05, t-test, 1 sided

3. Primary Outcome: Serum Sclerotin Levels
Description: Sclerostin has been proposed as the check-point where physical activity (PA) acts to modulate bone metabolism.
Time Frame: Baseline - W4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | No Additional Physical Exercise
Number analyzed (Participants) | 33
pmol/L
  Sclerostin, Baseline | 36.76 (9.68)
  Sclerostin, W4 | 37.30 (9.24)
Statistical Analysis 1: Comparison: No Additional Physical Exercise; Test type: Other; p = 0.05, t-test, 1 sided

4. Primary Outcome: Sclerostin
Description: Sclerostin has been proposed as the check-point where PA acts to modulate bone metabolism.
Time Frame: Week 4 - Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Physical Exercise
Number analyzed (Participants) | 33
pmol/L
  Sclerostin, W4 | 37.30 (9.24)
  Sclerostin, W12 | 33.96 (7.29)
Statistical Analysis 1: Comparison: Physical Exercise; Test type: Other; p = 0.05, t-test, 1 sided

5. Primary Outcome: Variation in Serum Carboxy-terminal Telopeptide of Collagen Type I (sCTX)
Description: Serum carboxy-terminal telopeptide of collagen type I (sCTX) is one of the most sensitive and specific bone resorption markers of osteoclast-mediated collagen degradation
Time Frame: Baseline - Week 4
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Control/Exercise Training: Usual care and no additional physical exercise
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
ng/mL
  sCTX baseline | 0.52 (0.13)
  sCTX, W4 | 0.53 (0.14)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

6. Primary Outcome: Variation of Serum Carboxy Terminal Telopeptide of Collagen Type I (sCTX)
Description: Serum carboxy terminal telopeptide of collagen type I (sCTX) is one of the most sensitive and specific bone resorption markers of osteoclast-mediated collagen degradation.
Time Frame: Week 4 - Week 12
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Control/Exercise Training: The exercise program was performed at C.U.R.I.A.Mo. Healthy Lifestyle Institute of Perugia University.
  The program provided 24 exercise sessions supervised by 2 physical education instructors and 2 medical researchers with a maximum attendance of 5 patient/group and carried out twice a week for three months.
  Each session lasted approximately 45 minutes divided into 15 minutes of cardiovascular activity performed using various ergometers and 30 minutes of weight-bearing endurance activities, resistance training and other exercise to develop balance and prevent falls, organized according to circuit training methodology.
  The great part of the exercise included in the program aim to provide variably strains (compression, bending, twisting) distributed across an higher surface of the femoral neck, to produce a maximal osteogenic response.
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
ng/mL
  sCTX, W4 | 0.53 (0.14)
  sCTX, W12 | 0.56 (0.15)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

7. Primary Outcome: Variation in Circulating Osteoprogenitor Cells (OPCs)
Description: Measurements of circulating OPCs with stem cell characteristics (CD34+) and express bone-specific proteins such as alkaline phosphatase (AP +) and osteocalcin (OCN +).
Time Frame: Baseline - Week 4
Measure: Mean (Standard Deviation); unit: cells/ml
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
cells/ml
  OCN+/CD34+ baseline | 1304.94 (782.79)
  OCN+/CD34+, W4 | 1393.92 (687.76)
  OCN+/AP+ baseline | 4485.21 (1690.12)
  OCN+/AP+, W4 | 4512.60 (1658.76)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

8. Primary Outcome: Variation in Circulating Osteoprogenitor Cells (OPCs).
Description: as for outcome 7
Time Frame: Week 4 - Week 12
Measure: Mean (Standard Deviation); unit: cells/ml
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
cells/ml
  OCN+/CD34+, W4 | 1393.92 (687.76)
  OCN+/CD34+, W12 | 2311.82 (1356.20)
  OCN+/AP+, W4 | 4512.60 (1658.76)
  OCN+/AP+, W12 | 5062.00 (1975.72)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

9. Secondary Outcome: Variation in Health-related Quality of Life (QoL)
Description: Health-related Quality of Life evaluated using the Quality of Life questionnaire of the European Foundation for Osteoporosis (QUALEFFO). The score ranges from 0, corresponding to the best QoL, to 100, corresponding to the worst QoL. Total score is the average value of 5 sub scores, corresponding to pain, physical function, mental function, social function and general health perception.
Time Frame: Baseline - Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
score on a scale
  Pain, Baseline | 22.59 (17.67)
  Pain, W4 | 21.97 (19.84)
  Physical function, Baseline | 9.89 (6.89)
  Physica function, W4 | 9.75 (6.52)
  Social function, Baseline | 24.38 (11.75)
  Social function, W4 | 23.77 (12.21)
  General health perception, Baseline | 43.23 (14.73)
  General health perception, W4 | 45.29 (14.12)
  Mental function, Baseline | 30.20 (10.89)
  Mental function, W4 | 30.09 (9.02)
  Total score, Baseline | 20.51 (7.06)
  Total score, W4 | 20.70 (7.11)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

10. Secondary Outcome: Variation in Health-related Quality of Life (QoL).
Description: as for outcome 9
Time Frame: Week 4 - Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control/Exercise Training
Number analyzed (Participants) | 33
score on a scale
  Pain, W4 | 21.97 (19.84)
  Physical function, W4 | 9.75 (6.52)
  Social function, W4 | 23.77 (12.21)
  General health perception, W4 | 45.29 (14.12)
  Mental function, W4 | 30.09 (9.02)
  Total score, W4 | 20.70 (7.11)
  Pain, W12 | 13.36 (12.45)
  Physical function, W12 | 8.13 (6.22)
  Social function, W12 | 22.10 (12.88)
  General health perception, W12 | 41.66 (14.47)
  Mental function, W12 | 28.55 (10.25)
  Total score, W12 | 18.55 (7.02)
Statistical Analysis 1: Comparison: Control/Exercise Training; Test type: Other; p = 0.05, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Control/Exercise Training
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Short duration of the observation (12 weeks). Small number of the sample. We did not provide any confirmation of the effects of the exercise program in terms of bone mineral density (BMD) or fracture risk.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No